CLINICAL TRIAL: NCT03170960
Title: A Phase 1b Dose-Escalation Study of Cabozantinib (XL184) Administered Alone or in Combination With Atezolizumab to Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of Cabozantinib Alone or in Combination With Atezolizumab to Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL184-021
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma; Renal Cell Carcinoma; Non-Small Cell Lung Cancer; Castration-resistant Prostate Cancer; Triple Negative Breast Cancer; Ovarian Cancer; Endometrial Cancer; Hepatocellular Carcinoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Colorectal Cancer; Head and Neck Cancer; Differentiated Thyroid Cancer; Lower Esophageal Cancer
Keywords: Kidney; Bladder; Renal pelvis; Ureter; Urethra; Cancer; Prostate; Castration-resistant; Lung; Breast; Ovarian; Endometrial; Liver; Stomach
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Neoplasms | interventions — cabozantinib; atezolizumab

STUDY DESIGN:
Intervention Model Description: Dose Escalation followed by Dose Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (25):
- Dose Escalation (Experimental): Subjects will accrue in cohorts of 3-6 subjects for evaluation of cabozantinib tablet dose of either 20 mg, 40 mg, and 60 mg orally qd in combination with standard dosing regimen of atezolizumab (1200 mg infusion q3w). A standard "3 plus 3" design will be utilized to determine a recommended combination dosing regimen for the Expansion Stage.
  Interventions: Drug: cabozantinib; Drug: atezolizumab
- Expansion Cohort 1 (Experimental): RCC subjects with clear cell histology who have not received prior systemic anticancer therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 2 (Experimental): UC subjects (including bladder, renal pelvis, ureter, urethra) who have progressed on or after platinum-containing chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 3 (Experimental): UC subjects (including bladder, renal pelvis, ureter, urethra) who are ineligible for cisplatin-based chemotherapy and have not received prior systemic chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 4 (Experimental): UC subjects (including bladder, renal pelvis, ureter, urethra) eligible for cisplatin-based chemotherapy and have not received prior systemic chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 5 (Experimental): UC subjects (including renal pelvis, ureter, urinary bladder, urethra) who have radiographically progressed on or after one prior immune check-point inhibitor (ICI) (anti-PD1 or anti-PD-L1) therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 6 (Experimental): CRPC subjects who have radiographically progressed in soft tissue on or after enzalutamide and/or abiraterone acetate for metastatic disease.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 7 (Experimental): Stage IV non-squamous NSCLC subjects who have radiographically progressed on or after treatment with one prior immune checkpoint inhibitor (ICI) (anti-PD-1 or anti-PD-L1) therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 8 (Experimental): Stage IV non-squamous NSCLC subjects with positive PD-L1 expression and without prior systemic anticancer therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 9 (Experimental): Stage IV nonsquamous NSCLC subjects with sensitizing EGFR mutation who have radiographically progressed during or following prior treatment with an EGFR-targeting TKI. Prior treatment with ICIs (anti-PD1 or anti-PD-L1) is allowed if given in combination with chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 10 (Experimental): RCC subjects with non-clear cell histology who have had up to one prior VEGFR-targeting TKI therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 11 (Experimental): TNBC subjects who have radiographically progressed during or following treatment with at least one prior systemic anticancer therapy. Prior treatment with ICIs (anti-PD1 or anti-PD-L1) is allowed if given in combination with chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 12 (Experimental): OC subjects (including primary peritoneal cancer and fallopian tube cancer) who have platinum-resistant or refractory disease who have had up to two lines of prior systemic anticancer therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 13 (Experimental): EC subjects (serous or endometrioid histology) who have radiographically progressed during or following treatment with at least one prior systemic anticancer therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 14 (Experimental): HCC subjects (Child-Pugh score A) who have not received prior systemic anticancer therapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 15 (Experimental): GC/GEJC/LEC subjects who have radiographically progressed during or following platinum-containing or fluoropyrimidine-containing chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 16 (Experimental): CRC subjects who have radiographically progressed during or following systemic chemotherapy that contained fluoropyrimidine in combination with oxaliplatin or irinotecan.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 17 (Experimental): H&N cancer subjects who have radiographically progressed during or following prior platinum-containing chemotherapy. Prior treatment with ICIs (anti-PD1 or anti-PD-L1) is allowed if given in combination with chemotherapy.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 18 (Experimental): DTC subjects (follicular, papillary, and poorly differentiated histologies) who are radioactive iodine (RAI) refractory or deemed ineligible for treatment with RAI.
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 19 (SAC) (Experimental): UC subjects (including renal pelvis, ureter, urinary bladder, urethra) who have radiographically progressed on or after one prior ICI (anti-PD-1 or anti-PD-L1). Subjects may be allowed to receive combination therapy at the Cohort Review Committee recommended dose following radiographic disease progression.
  Interventions: Drug: cabozantinib
- Expansion Cohort 20 (SAC) (Experimental): Stage IV non-squamous NSCLC subjects who have radiographically progressed on or after treatment with one prior ICI (anti-PD-1 or anti-PD-L1). Subjects may be allowed to receive combination therapy at the Cohort Review Committee recommended dose following radiographic disease progression.
  Interventions: Drug: cabozantinib
- Expansion Cohort 21 (SAC) (Experimental): Metastatic CRPC (mCRPC) subjects who have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features who have had prior treatment with one, and only one, novel hormonal therapy (NHT) (eg, abiraterone, enzalutamide, apalutamide, daralutamide) for CSPC, mCRPC, or non-metastatic CRPC. Subjects may be allowed to receive combination therapy at the Cohort Review Committee recommended dose following radiographic disease progression.
  Interventions: Drug: cabozantinib
- Expansion Cohort 22 (SAA) (Experimental): Metastatic CRPC (mCRPC) subjects who have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features who have had prior treatment with one, and only one, novel hormonal therapy (NHT) (eg, abiraterone, enzalutamide, apalutamide, daralutamide) for CSPC, mCRPC, or non-metastatic CRPC. Subjects may be allowed to receive combination therapy at the Cohort Review Committee recommended dose following radiographic disease progression.
  Interventions: Drug: atezolizumab
- Expansion Cohort 23 (Experimental): Metastatic CRPC (mCRPC) subjects who have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features who have had prior treatment with one, and only one, novel hormonal therapy (NHT) (eg, abiraterone, enzalutamide, apalutamide, daralutamide) for CSPC, mCRPC, or non-metastatic CRPC
  Interventions: Drug: atezolizumab; Drug: cabozantinib
- Expansion Cohort 24 (Experimental): Metastatic CRPC (mCRPC) subjects who have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features who have had prior treatment with at least one NHT and have received docetaxel for mCRPC
  Interventions: Drug: atezolizumab; Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — Supplied as 60-mg and 20-mg tablets; administered orally daily at dose levels of 20 mg, 40 mg, or 60 mg.
  Other Names: Cabometyx; XL184
  Arms: Dose Escalation
Drug: atezolizumab — Supplied as 1200-mg vials; administered as an IV infusion once every 3 weeks (q3w).
  Other Names: Tecentriq
  Arms: Dose Escalation; Expansion Cohort 1; Expansion Cohort 10; Expansion Cohort 11; Expansion Cohort 12; Expansion Cohort 13; Expansion Cohort 14; Expansion Cohort 15; Expansion Cohort 16; Expansion Cohort 17; Expansion Cohort 18; Expansion Cohort 2; Expansion Cohort 22 (SAA); Expansion Cohort 23; Expansion Cohort 24; Expansion Cohort 3; Expansion Cohort 4; Expansion Cohort 5; Expansion Cohort 6; Expansion Cohort 7; Expansion Cohort 8; Expansion Cohort 9
Drug: cabozantinib — Supplied as 60-mg and 20-mg tablets; administered orally daily at the Cohort Review Committee-determined recommended dose from the Dose Escalation Stage
  Other Names: Cabometyx; XL184
  Arms: Expansion Cohort 1; Expansion Cohort 10; Expansion Cohort 11; Expansion Cohort 12; Expansion Cohort 13; Expansion Cohort 14; Expansion Cohort 15; Expansion Cohort 16; Expansion Cohort 17; Expansion Cohort 18; Expansion Cohort 2; Expansion Cohort 23; Expansion Cohort 24; Expansion Cohort 3; Expansion Cohort 4; Expansion Cohort 5; Expansion Cohort 6; Expansion Cohort 7; Expansion Cohort 8; Expansion Cohort 9
Drug: cabozantinib — Supplied as 60-mg and 20-mg tablets; administered orally daily at 60 mg qd
  Other Names: Cabometyx; XL184
  Arms: Expansion Cohort 19 (SAC); Expansion Cohort 20 (SAC); Expansion Cohort 21 (SAC)

SUMMARY:
This is a multicenter Phase 1b, open-label study to assess safety, tolerability, preliminary efficacy, and pharmacokinetics (PK) of cabozantinib taken in combination with atezolizumab in subjects with multiple tumor types, including advanced urothelial carcinoma (UC) (including bladder, renal pelvis, ureter, urethra), renal cell carcinoma (RCC), castration-resistant prostate cancer (CRPC), non-small-cell lung cancer (NSCLC), triple negative breast cancer (TNBC), ovarian cancer (OC), endometrial cancer (EC), hepatocellular cancer (HCC), gastric cancer/gastroesophageal junction cancer/lower esophageal cancer (GC/GEJC/LEC), colorectal cancer (CRC), head and neck (H&N) cancer, and differentiated thyroid cancer (DTC). The study consists of two stages: in the Dose Escalation Stage, an appropriate recommended cabozantinib dose for the combination with standard dosing regimen of atezolizumab will be established; in the Expansion Stage, tumor-specific cohorts will be enrolled in order to further evaluate the safety and efficacy of the combination treatment in these tumor indications. Three exploratory single-agent cabozantinib (SAC) cohorts may also be enrolled with UC, NSCLC, or CRPC subjects. One exploratory single-agent atezolizumab (SAA) cohort may also be enrolled with CRPC subjects. Subjects enrolled in the SAC cohorts and SAA cohort may receive combination treatment with both cabozantinib and atezolizumab after they experience radiographic progressive disease per the Investigator per RECIST 1.1. Due to the nature of this study design, some tumor cohorts may complete enrollment earlier than others.

DETAILED DESCRIPTION:
* Dose Escalation Stage: to determine the schedule and maximum tolerated dose (MTD) and/or recommended Expansion Stage dose of cabozantinib when taken in combination with a standard dosing regimen of atezolizumab (1200 mg infusion, once every 3 weeks).
* Expansion Stage: to determine the preliminary efficacy (objective response rate [ORR] per RECIST 1.1) and safety of the recommended combination dose of cabozantinib with atezolizumab in eighteen tumor-specific cohorts including subjects with advanced UC, RCC, CRPC, NSCLC, TNBC, OC, EC, HCC, GC/GEJC/LEC, CRC, H&N, and DTC.
* Exploratory SAC Cohorts: Descriptive efficacy, safety, PK, and biomarker analyses of single-agent cabozantinib in UC, NSCLC, and CRPC subjects. Descriptive efficacy and safety analyses of combination therapy after progression on single-agent therapy
* Exploratory SAA Cohort: Descriptive efficacy, safety, PK, and biomarker analyses of single-agent atezolizumab in CRPC subjects. Descriptive efficacy and safety analyses of combination therapy after progression on single-agent therapy

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically and radiologically confirmed solid tumor that is inoperable, locally advanced, metastatic, or recurrent:

   * Dose-Escalation Stage:

     * Subjects with UC (including renal pelvis, ureter, bladder, urethra) after prior platinum-based therapy, or
     * Subjects with RCC (clear cell, non-clear cell histology) with or without prior systemic anticancer therapy
   * Expansion Stage:

     * Inoperable locally advanced or metastatic solid tumor (UC, RCC, CRPC, NSCLC, TNBC, OC, EC, HCC, GC/GEJC/LEC, CRC, H&N cancer, and DTC as outlined above)
2. Measurable disease per RECIST 1.1 as determined by the investigator.
3. Tumor tissue material available (archival or recent tumor biopsy)
4. Recovery to baseline or ≤ Grade 1 CTCAE v4 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
5. Age eighteen years or older on the day of consent.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Adequate organ and marrow function.
8. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception.
9. Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

1. Prior treatment with cabozantinib or immune checkpoint inhibitors including anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy except in Expansion Cohorts 5, 7, 9, 11, 17, 19 and 20. Other restrictions regarding prior therapy may apply.
2. Known brain metastases or cranial epidural disease unless adequately treated and stable for at least 4 weeks before first dose of study treatment.
3. Concomitant anticoagulation with oral anticoagulants.
4. Subject is receiving systemic steroid therapy (>10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to first dose of study treatment.
5. Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.
6. The subject has uncontrolled, significant intercurrent or recent illness, including, but not limited to, an active or history of autoimmune disease or immune deficiency; idiopathic pulmonary fibrosis, organizing pneumonia, pneumonitis; active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV), AIDS-related illness, acute or chronic hepatitis B or C infection, positive test for tuberculosis, moderate to severe hepatic impairment (Child-Pugh B or C).
7. Pregnant or lactating females.
8. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
9. Diagnosis of another malignancy within 2 years before first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: MTD/Recommended Dose | Up to Day 21
  To determine the maximum tolerated dose (MTD) and/or recommended dose and schedule for the subsequent Expansion Stage of daily oral administration of cabozantinib in subjects with solid tumors when taken in combination with atezolizumab.
Dose Expansion: ORR | Up to a maximum of 59 months
  To evaluate preliminary efficacy by estimating the Objective Response Rate (ORR) as assessed by the Investigator per RECIST 1.1.

SECONDARY OUTCOMES:
Incidence and severity of nonserious AEs and SAEs (Safety) | From first dose to 30 days following last dose (up to a maximum of 59 months)
  To assess safety for the combination therapy through the evaluation of incidence and severity of nonserious adverse events (AEs) and serious adverse events (SAEs), including immune-related adverse events (irAEs) and adverse events of special interest (AESIs).

CONTACTS AND LOCATIONS:
Locations (124):
- United States (57):
  - Exelixis Clinical Site #53, Gilbert, Arizona
  - Exelixis Clinical Site #18, Phoenix, Arizona
  - Exelixis Clinical Site #1, Duarte, California
  - Exelixis Clinical Site #20, La Jolla, California
  - Exelixis Clinical Site #46, Los Angeles, California
  - Exelixis Clinical Site #51, Newport Beach, California
  - Exelixis Clinical Site #62, Santa Monica, California
  - Exelixis Clinical Site #21, Stanford, California
  - Exelixis Clinical Site #34, Denver, Colorado
  - Exelixis Clinical Site #50, Denver, Colorado
  - Exelixis Clinical Site #42, New Haven, Connecticut
  - Exelixis Clinical Site #48, Washington D.C., District of Columbia
  - Exelixis Clinical Site #16, Jacksonville, Florida
  - Exelixis Clinical Site #76, Tampa, Florida
  - Exelixis Clinical Site #60, Atlanta, Georgia
  - Exelixis Clinical Site #79, Atlanta, Georgia
  - Exelixis Clinical Site #32, Harvey, Illinois
  - Exelixis Clinical Site #23, Fairway, Kansas
  - Exelixis Clinical Site #57, Lexington, Kentucky
  - Exelixis Clinical Site #24, New Orleans, Louisiana
  - Exelixis Clinical Site #10, Boston, Massachusetts
  - Exelixis Clinical Site #3, Detroit, Michigan
  - Exelixis Clinical Site #17, Rochester, Minnesota
  - Exelixis Clinical Site #65, Bolivar, Missouri
  - Exelixis Clinical Site #43, Kansas City, Missouri
  - Exelixis Clinical Site #35, Omaha, Nebraska
  - Exelixis Clinical Site #59, Omaha, Nebraska
  - Exelixis Clinical Site #61, Las Vegas, Nevada
  - Exelixis Clinical Site #38, Camden, New Jersey
  - Exelixis Clinical Site #27, East Brunswick, New Jersey
  - Exelixis Clinical Site #31, New Brunswick, New Jersey
  - Exelixis Clinical Site #40, East Setauket, New York
  - Exelixis Clinical Site #11, New York, New York
  - Exelixis Clinical Site #37, The Bronx, New York
  - Exelixis Clinical Site #67, Cleveland, Ohio
  - Exelixis Clinical Site #49, Columbus, Ohio
  - Exelixis Clinical Site #64, Kettering, Ohio
  - Exelixis Clinical Site #71, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #6, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #102, Portland, Oregon
  - Exelixis Clinical Site #45, Portland, Oregon
  - Exelixis Clinical Site #41, Bethlehem, Pennsylvania
  - Exelixis Clinical Site #15, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #55, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #66, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #95, Charleston, South Carolina
  - Exelixis Clinical Site #13, Dallas, Texas
  - Exelixis Clinical Site #26, Dallas, Texas
  - Exelixis Clinical Site #114, Fort Worth, Texas
  - Exelixis Clinical Site #29, Houston, Texas
  - Exelixis Clinical Site #39, Houston, Texas
  - Exelixis Clinical Site #44, Houston, Texas
  - Exelixis Clinical Site #33, Lubbock, Texas
  - Exelixis Clinical Site #63, San Antonio, Texas
  - Exelixis Clinical Site #2, Salt Lake City, Utah
  - Exelixis Clinical Site #30, Blacksburg, Virginia
  - Exelixis Clinical Site #14, Charlottesville, Virginia
- Australia (6):
  - Exelixis Clinical Site #98, Albury, New South Wales
  - Exelixis Clinical Site #101, Camperdown, New South Wales
  - Exelixis Clinical Site #115, Gosford, New South Wales
  - Exelixis Clinical Site #112, North Ryde, New South Wales
  - Exelixis Clinical Site #123, Randwick, New South Wales
  - Exelixis Clinical Site #99, St Albans, Victoria
- Belgium (2):
  - Exelixis Clinical Site #52, Ghent
  - Exelixis Clinical Site #54, Leuven
- France (19):
  - Exelixis Clinical Site #88, La Roche-sur-Yon, Cedex 9
  - Exelixis Clinical Site #8, Villejuif, Cedex
  - Exelixis Clinical Site #92, Bordeaux
  - Exelixis Clinical Site #93, Brest
  - Exelixis Clinical Site #87, Caen
  - Exelixis Clinical Site #69, Le Mans
  - Exelixis Clinical Site #97, Lille
  - Exelixis Clinical Site #89, Lyon
  - Exelixis Clinical Site #109, Marseille
  - Exelixis Clinical Site #104, Nice
  - Exelixis Clinical Site #80, Nîmes
  - Exelixis Clinical Site #78, Paris
  - Exelixis Clinical Site #7, Paris
  - Exelixis Clinical Site #68, Paris
  - Exelixis Clinical Site #72, Paris
  - Exelixis Clinical Site #82, Saint-Grégoire
  - Exelixis Clinical Site #119, Strasbourg
  - Exelixis Clinical Site #107, Suresnes
  - Exelixis Clinical Site #105, Vandœuvre-lès-Nancy
- Germany (2):
  - Exelixis Clinical Site #56, Düsseldorf, North Rhine-Westphalia
  - Exelixis Clinical Site #36, Tübingen
- Italy (9):
  - Exelixis Clinical Site #84, Meldola, FC
  - Exelixis Clinical Site #47, Rozzano, Milano
  - Exelixis Clinical Site #108, Milan
  - Exelixis Clinical Site #103, Milan
  - Exelixis Clinical Site #25, Milan
  - Exelixis Clinical Site #4, Milan
  - Exelixis Clinical Site #85, Napoli
  - Exelixis Clinical Site #121, Pavia
  - Exelixis Clinical Site #110, Roma
- Exelixis Clinical Site #12, Nijmegen, Gelderland, Netherlands
- Spain (24):
  - Exelixis Clinical Site #74, Santiago de Compostela, A Coruña
  - Exelixis Clinical Site #91, Elche, Alicante
  - Exelixis Clinical Site #70, Palma de Mallorca, Balearic Islands
  - Exelixis Clinical Site #113, Badalona, Barcelona
  - Exelixis Clinical Site #116, Sabadell, Barcelona
  - Exelixis Clinical Site #96, Jeréz de La Frontera, Cádiz
  - Exelixis Clinical Site #90, Pamplona, Navarre
  - Exelixis Clinical Site #94, Oviedo, Principality of Asturias
  - Exelixis Clinical Site #117, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Exelixis Clinical Site #75, Barcelona
  - Exelixis Clinical Site #58, Barcelona
  - Exelixis Clinical Site #83, Barcelona
  - Exelixis Clinical Site #86, Barcelona
  - Exelixis Clinical Site #28, Barcelona
  - Exelixis Clinical Site #9, Barcelona
  - Exelixis Clinical Site #73, Barcelona
  - Exelixis Clinical Site #118, Girona
  - Exelixis Clinical Site #77, Madrid
  - Exelixis Clinical Site #106, Madrid
  - Exelixis Clinical Site #111, Madrid
  - Exelixis Clinical Site #22, Madrid
  - Exelixis Clinical Site #5, Madrid
  - Exelixis Clinical Site #81, Madrid
  - Exelixis Clinical Site #100, Málaga
- United Kingdom (4):
  - Exelixis Clinical Site #122, Middlesex, England
  - Exelixis Clinical Site #120, Preston, England
  - Exelixis Clinical Site #124, Cardiff, Wales
  - Exelixis Clinical Site #19, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pal SK, Loriot Y, Necchi A, Singh P, Castellano D, Pagliaro L, Suarez C, McGregor BA, Vaishampayan UN, Hauke RJ, Powles T, Van Herpen CML, Courtney KD, Dreicer R, Sudhagoni R, Schwickart M, Andrianova S, Agarwal N. COSMIC-021 Phase Ib Study of Cabozantinib Plus Atezolizumab: Results from the Locally Advanced or Metastatic Urothelial Carcinoma Cohorts. J Clin Oncol. 2025 May 10;43(14):1650-1662. doi: 10.1200/JCO-24-01675. Epub 2025 Feb 18. PMID 39965176
- [Derived] Li D, Loriot Y, Burgoyne AM, Cleary JM, Santoro A, Lin D, Aix SP, Garrido-Laguna I, Sudhagoni R, Guo X, Andrianova S, Paulson S. Cabozantinib plus atezolizumab in previously untreated advanced hepatocellular carcinoma and previously treated gastric cancer and gastroesophageal junction adenocarcinoma: results from two expansion cohorts of a multicentre, open-label, phase 1b trial (COSMIC-021). EClinicalMedicine. 2023 Dec 21;67:102376. doi: 10.1016/j.eclinm.2023.102376. eCollection 2024 Jan. PMID 38204489
- [Derived] Agarwal N, McGregor B, Maughan BL, Dorff TB, Kelly W, Fang B, McKay RR, Singh P, Pagliaro L, Dreicer R, Srinivas S, Loriot Y, Vaishampayan U, Goel S, Curran D, Panneerselvam A, Schwickart M, Choueiri TK, Pal S. Cabozantinib in combination with atezolizumab in patients with metastatic castration-resistant prostate cancer: results from an expansion cohort of a multicentre, open-label, phase 1b trial (COSMIC-021). Lancet Oncol. 2022 Jul;23(7):899-909. doi: 10.1016/S1470-2045(22)00278-9. Epub 2022 Jun 9. PMID 35690072
- [Derived] Pal SK, McGregor B, Suarez C, Tsao CK, Kelly W, Vaishampayan U, Pagliaro L, Maughan BL, Loriot Y, Castellano D, Srinivas S, McKay RR, Dreicer R, Hutson T, Dubey S, Werneke S, Panneerselvam A, Curran D, Scheffold C, Choueiri TK, Agarwal N. Cabozantinib in Combination With Atezolizumab for Advanced Renal Cell Carcinoma: Results From the COSMIC-021 Study. J Clin Oncol. 2021 Nov 20;39(33):3725-3736. doi: 10.1200/JCO.21.00939. Epub 2021 Sep 7. PMID 34491815